CLINICAL TRIAL: NCT02968212
Title: Phase 2 Study of Clofazimine for the Treatment of Pulmonary Mycobacterium Avium Disease
Brief Title: Clofazimine in the Treatment of Pulmonary Mycobacterium Avium Complex (MAC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Jewish Health (Other); The University of Texas Health Science Center at Tyler (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Chicago (Other); Temple University (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Kevin Winthrop, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FD-R-5401
Record Dates: First submitted 2016-11-10; First posted 2016-11-18 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Mycobacterium Avium Complex
Keywords: Mycobacterium avium Complex; Clofazimine
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection | interventions — Clofazimine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- clofazimine (Experimental): Participants receive lamprene
  Interventions: Drug: Clofazimine
- sugar pill (Placebo Comparator): Participants receive placebo
  Interventions: Other: sugar pill

INTERVENTIONS:
Drug: Clofazimine — All participants in the experimental/treatment arm on this protocol will take a loading dose of 200 mg daily in soft capsule form of clofazimine for 16 weeks, dropping to 100 mg daily for the next 8 weeks.
  Other Names: Lamprene
  Arms: clofazimine
Other: sugar pill — All participants in the placebo arm on this protocol will take placebo in soft capsule form daily dropping to a smaller dose after 16 weeks to mirror the treatment arm dosing.
  Other Names: placebo
  Arms: sugar pill

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness and safety of clofazimine when used to treat Mycobacteria avium complex (MAC) lung disease.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Clofazimine is an orphan antibiotic drug that is no longer available through pharmacies in the United States. It is approved for the treatment of Mycobacterium leprae (leprosy) infections. Clofazimine has been used for many years off-label against other Mycobacterium, including Mycobacteria avium complex (MAC) lung disease, an increasingly prevalent infection in older Americans. The U.S. Food and Drug Administration currently oversees clofazimine use to treat MAC lung disease through a special investigational drug access program. However, to date, there is little understanding of the benefits and risks of clofazimine when used to treat MAC lung disease. Accordingly, the investigators have developed a randomized, placebo-controlled clinical trial to assess the clinical efficacy and safety of clofazimine. To be eligible, participants must have MAC lung disease, positive sputum cultures for MAC, and not currently taking antibiotics for MAC. Eligible participants (102 total enrolled) will be randomly given either clofazimine or placebo for 6 months, and followed closely by their treating physician. The percentage of participants who become culture negative in each group will be compared, as it is suspected that participants treated with clofazimine will be more likely to become culture negative. The safety of clofazimine will be measured as well as other potential benefits of the therapy including changes in lung function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 positive MAC sputum cultures in the last 12 months with at least one obtained within 12 weeks prior to randomization
* Meet ATS/IDSA 2007 pulmonary disease criteria
* Adult males and females age 18 or over
* Ability to provide informed consent for the use of study drug

Exclusion Criteria:

* Any patient who is unwilling or unable to provide consent or to comply with this protocol
* Cavitary NTM disease
* Patients who are currently taking or within the prior 12 weeks received any of the following: bedaquiline, or any component of ATS/IDSA multi-drug recommended therapy (macrolide, ethambutol, rifampin) for MAC
* Current usage of inhaled amikacin, tobramycin, or gentamicin
* In the judgment of the investigator, the patient is not a candidate for observation (e.g. severe symptoms, extensive disease burden) but rather should be treated with standard multi-drug therapy
* Prior use of clofazimine that has resulted in an allergy to clofazimine or a severe adverse reaction
* Current usage of medications associated with QT prolongation (see Appendix C for full list of prohibited concomitant medications)
* Corrected QT (QTc) interval on electrocardiogram (ECG) > 470 ms for females or 450 ms for males, calculated using Fridericia's formula60,61
* Advanced lung disease (FEV<30%)
* HIV
* Active pulmonary tuberculosis requiring treatment at screening
* Active pulmonary malignancy or chemotherapy or radiation within 1 year of screening
* Use of chronic systemic corticosteroids at doses of 15 mg/day for more than 12 weeks
* Prior lung or other solid organ transplant
* Pregnancy, or breastfeeding that will continue during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline sputum culture at 24 weeks | Sputum examined for culture change from Baseline at 24 weeks
  sputum will be processed for acid fast bacilli stain/acid fast bacterial culture. A semi-quantitative assessment will be made by colony count for patients.

SECONDARY OUTCOMES:
Change from Baseline 6 Minute Walk Test at 24 weeks | 6 Minute Walk Test results examined for change from Baseline at 24 weeks
  Walking distance achieved in 6 minutes is assessed
Change from Baseline PROMIS Fatigue 7a short form questionnaire at 24 weeks | PROMIS Fatigue 7a short form results examined for change from Baseline at 24 weeks
  Self-administered questionnaire assessing a range of self-reported symptoms over the past seven days, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities.
Change from Baseline Quality of Life-Bronchiectasis (QOL-B) with NTM module at 24 weeks | QOL-B results examined for change from Baseline at 24 weeks
  Self-administered questionnaire measuring 8 separate domains: Physical Functioning, Role Functioning, Vitality, Emotional Functioning, Social Functioning, Treatment Burden, Health Perceptions, and Respiratory Symptoms.
Change from Baseline CT scan at 24 weeks | CT scan examined for change from Baseline at 24 weeks
  CT scans will be computationally evaluated using custom software to provide volumetric assessment of NTM-associated abnormalities.
Change from Baseline semi-quantitative sputum acid fast smear culture at 24 weeks | semi-quantitative sputum acid fast smear culture examined for change from Baseline at 24 weeks
  sputum will be processed for acid fast bacilli stain/acid fast bacterial culture. A semi-quantitative assessment will be made by colony count for patients.
Change from Baseline Spirometry at 24 weeks | Spirometry with FEV1/FVC ratio examined for change from Baseline at 24 weeks
  Mean change in pulmonary function parameters as measured by %predicted FEV1 and FVC
Change from Baseline Erythrocyte Sedimentation Rate at 24 weeks | Erythrocyte Sedimentation Rate examined for change from Baseline at 24 weeks
  Detecting change in Inflammatory markers
Change from Baseline C-Reactive Protein levels at 24 weeks | C-Reactive Protein levels examined for change from Baseline at 24 weeks
  Detecting change in Inflammatory markers
Number of Adverse Events | Number of Patient-reported and Investigator-reported Adverse Events at 24 weeks
  Comparison of experienced adverse events between the two study groups
Change from Baseline QT interval at 24 weeks | QT interval examined for change from Baseline at 24 weeks
  A 12-lead ECG will be conducted, and the QT interval calculated using Fridericia's formula: QTC = QT / RR 1/3
Change from Baseline blood serum chemistry at week 24 | blood serum chemistry examined for change from Baseline at 24 weeks
  Detecting changes in liver ALT and AST levels
Change from Baseline complete blood count at week 24 | complete blood count examined for change from Baseline at 24 weeks
  Detecting changes in complete blood count
Change from Baseline Minimal Inhibitory Concentration of MAC isolates in vitro at week 24 | Minimal Inhibitory Concentration of MAC isolates in vitro examined for change from Baseline at 24 weeks
  Detecting change in MAC isolates sensitivity to clofazimine

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Winthrop, MD, Principal Investigator — Oregon Health and Science University
Locations (7):
- United States (7):
  - National Jewish Health, Denver, Colorado
  - University of South Florida, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Louisiana State University, Baton Rouge, Louisiana
  - National Heart, Lung and Blood Institute, Bethesda, Maryland
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Health Science Center, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No